CLINICAL TRIAL: NCT05870553
Title: A Prospective, Randomized, Single-blinded (Evaluator), Parallel, Multi-center, Phase 3 Trial in Bowel Preparation for Colonoscopy.
Brief Title: A Phase 3 Trial in Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP0301
Record Dates: First submitted 2023-04-21; First posted 2023-05-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CTP0301-A (Experimental): Subjects who are randomized into this group will take CTP0301-A from the evening before colonoscopy to the morning of colonoscopy.
  Interventions: Drug: CTP0301-A
- CTP0301-B (Experimental): Subjects who are randomized into this group will take CTP0301-B before the morning of colonoscopy.
  Interventions: Drug: CTP0301-B
- Cool prep (Active Comparator): Subjects who are randomized into this group will take Cool prep from the evening before colonoscopy to the morning of colonoscopy.
  Interventions: Drug: Cool prep

INTERVENTIONS:
Drug: CTP0301-A — Bowel Preparation
  Other Names: PEG 3350
  Arms: CTP0301-A
Drug: CTP0301-B — Bowel Preparation
  Other Names: PEG 3350
  Arms: CTP0301-B
Drug: Cool prep — Bowel Preparation
  Other Names: PEG 3350
  Arms: Cool prep

SUMMARY:
This is a prospective randomized study compared with active control arm. The investigators compare the colon cleansing in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients and inpatients aged: ≥19
* A prospective colonoscopy person
* Written informed consent to participate in the trial

Exclusion Criteria:

* Patients with past history of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease.
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, subtotal colectomy, abdominoperineal resection, defunctioning colostomy.
* Pregnant women or pregnant women or pregnant women
* Severe heart disease (cardiac failure (NYHA class 3 and 4))
* Acute coronary artery disease within 24 weeks before screening (an unstable angina pectoris, acute myocardial infarction), clinically significant arrhythmia, hypertrophic obstruction Cardiomyopathy, valvular disease, aortic and peripheral vascular diseases.
* People who have hypersensitivity or allergies to clinical trial drug components.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Number of Patients With Successful Bowel Cleansing (Overall Colon) | 1 day of scheduled colonoscopy
  The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e. all mucosa could be visualized) and C and D are classified as unsuccessful.

SECONDARY OUTCOMES:
Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens) | 1 day of scheduled colonoscopy
  The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). Highly effective cleansing in the colon ascendens corresponded to scores 3 (Good) or 4 (Excellent) of the HCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No